CLINICAL TRIAL: NCT05542732
Title: Accuracy of CardioWatch 287-2 During Profound Hypoxia
Acronym: ACW2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corsano Health B.V. (Industry)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CIV-21-12-038447
Record Dates: First submitted 2022-09-09; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Hypoxia
Keywords: oxygen saturation; heart rate; respiratory rate; SpO2; wrist wearable; PPG; Corsano; CardioWatch 287-2; accuracy
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: A sample size of twelve subjects was planned in both the non-invasive study and invasive study, as recommended by the FDA Guidance for Industry and FDA Staff Pulse Oximeters - Premarket Notification Submissions [510(k)s]. Of these subjects, at least a minimum of 2 subjects or 15% of the analyzed population needed to have a dark skin pigmentation and at least 30 % of one gender is preferred.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental): Each participant wore one CW2 sensor attached to the back of the wrist with a wrist band. Additionally, each participant wore a reference pulse oximeter (Nellcor PM10) attached to the middle finger of the ipsilateral hand. This enabled the comparison of the paired results of the CW2 sensor and reference pulse oximeter equipment for SpO2 measurements at different oxygen saturation levels. Twelve subjects of the 24 participants received an arterial catheter in the contralateral radial artery for exvivo SaO2 determination by CO-oximetry and in order to define the final accuracy of CW2 for SpO2 measurement.
  Interventions: Device: CardioWatch 287-2

INTERVENTIONS:
Device: CardioWatch 287-2 — CardioWatch 287-2 (CW2 Test Device or CW2). This medical device is based on the precursor CardioWatch 287-1 approved by EU-MDR under number 20M00011CRT01, CW2 has two red, two infrared and two green LEDs, and two photosensors compared to its precursor.

SUMMARY:
In an individual's SpO2 range from 100 to 73 %, this study calibrates and evaluates the accuracy of SpO2 measurement by CW2 in comparison to reference pulse oximeter (Nellcor PM10) or CO-oximetry, Pulse rate (PR) and respiratory rate (RR) were calibrated based on the same Nellcor equipment and the frequency of end-tidal CO2 respectively.

DETAILED DESCRIPTION:
The study is designed in accordance with Medical electrical equipment - Part 2-61: Particular requirements for basic safety and essential performance of pulse oximeter equipment ISO 80601-2-61:2017, Corrected version 2018-02 and ISO 80601-2-55.

SpO2: Testing to confirm the accuracy of the SpO2 monitoring according to ISO 80601-2-61 Clause 201.12.1.101 201.12.1.101

RR Testing: Testing to confirm the accuracy of the respiration rate monitoring according to ISO 80601-2-55. Volunteers respirated spontaneously, no efforts were made to include all ranges of respiration during the study.

PR Testing: Testing to confirm the accuracy of the PR monitoring according to ISO 80601-2-61 Clause 201.12.1.104. No efforts were made to influence PRs of volunteers.

An accelerometer and PPG filters are built in CW2 in order to form the basis to exclude non-eligible test results.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy non-disabled subjects with American Society of Anesthesiologists health score (ASA) of 1 or 2.
2. The subject is aged ≥18 and ≤ 65 years.
3. The subject is not intellectual disabled, and has provided informed consent and is willing to comply with the study procedures.

Exclusion Criteria:

1. Heavy smokers or individuals exposed to high levels of carbon monoxide that result in elevated carboxyhemoglobin levels.
2. Individuals subject to conditions that result in elevated levels of methemoglobin
3. Individuals with hypoxia (SpO2 < 95 % at 21 % of oxygen)
4. Severe claustrophobia
5. Subject is known with altitude disease
6. The subject is obese (BMI ≥ 31 kg/m2).
7. The subject has a known history of moderate to severe heart disease, lung disease, kidney or liver disease.
8. The subject is diagnosed with moderate to severe asthma.
9. The subject is known with a hemoglobinopathy or history of anemia, e.g. sickle cell anemia, thalassemia, ... who, in the opinion of the investigator, would make them unsuitable for study participation.
10. The subject has any other serious systemic illness.
11. Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators would interfere with the sensors working correctly.
12. The subject has a history of fainting or vasovagal response.
13. The subject has a history of sensitivity or allergy to local anesthetics or disinfectants.
14. The subject has a diagnosis of Raynaud's disease.
15. The subject has unacceptable collateral circulation based on exam by the investigator.
16. The subject is pregnant, lactating or trying to get pregnant.
17. The subject is unable or unwilling to provide informed consent or is unable or unwilling to comply with study procedures.
18. The subject has any other condition, which in the opinion of the investigators would make the subject unsuitable for the study.
19. The subject refuses to remove nail-vanish.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-04 (Actual); Primary Completion 2022-06-18 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Pulse Oximetry | 1 hour
  SpO2
Pulse rate | 1 hour
  Heart rate in beats per minutes
Respiratory rate | 1 hour
  In breaths per minutes

CONTACTS AND LOCATIONS:
Overall Officials: Raf de Jongh, MD, PhD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Complementair Medisch Centrum (CMC) Europe, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No